CLINICAL TRIAL: NCT03837808
Title: A Randomized Phase III Non-inferiority Study of Radiotherapy Plus Concurrent Nimotuzumab Versus Cisplatin in Stage II-III Nasopharyngeal Carcinoma
Brief Title: Radiotherapy Plus Concurrent Nimotuzumab or Cisplatin in Stage II-III Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-206
Record Dates: First submitted 2019-01-26; First posted 2019-02-12 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasm
Keywords: nimotuzumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasms | interventions — nimotuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab (Experimental): nimotuzumab 200mg/week in concurrent with IMRT
  Interventions: Drug: Nimotuzumab
- Cisplatin (Active Comparator): cisplatin 40mg/m2/week in concurrent with IMRT
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Nimotuzumab — nimotuzumab 200mg/week in concurrent with IMRT, d1,d8,d15,d22,d29,d36 of RT
  Arms: Nimotuzumab
Drug: Cisplatin — cisplatin 40mg/m2/week in concurrent with IMRT, d1,d8,d15,d22,d29,d36 of RT
  Arms: Cisplatin

SUMMARY:
This is a Phase III trial to study the effectiveness of nimotuzumab versus cisplatin combined with intensity-modulated radiation therapy (IMRT) in treating patients with stage II-III nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Scheme:

Eligible stage II and III NPC patients will first be stratified by institution, then randomized to 2 arms at 1:1 ratio.

- Arm Cisplatin: cisplatin 40mg/m2/week in concurrent with IMRT

- Arm nimotuzumab: nimotuzumab 200mg/week in concurrent with IMRT

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* histologically confirmed positive EGFR expression
* Stage II and III NPC patients（according to the 8th AJCC edition）
* Male and no pregnant female
* Age between 18-65
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <2.0×upper limit of normal (ULN)
* Adequate renal function: creatinine clearance ≥60 ml/min
* Satisfactory performance status: Karnofsky scale (KPS) > 70
* Without radiotherapy or chemotherapy
* Patients must give signed informed consent

Exclusion Criteria:

* Evidence of relapse or distant metastasis
* History of prior malignancy or previous treatment for NPC
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-02-11 (Estimated); Study Completion 2024-02-11 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRRFS) | 2 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant Metastasis-Free Survival (DMFS) | 2 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Number of participants with adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China